CLINICAL TRIAL: NCT06224335
Title: Femfit® and an Innovative Pad Test to Assess Pelvic Floor Muscle Activation During Physical Activity in Sportwoman with and Without SUI - a Pilot Study
Brief Title: Measurement of Intravaginal and Intra-abdominal Pressure and Pad Test During Sports Activities (SPORTVAGPRES)
Acronym: SPORTVAGPRES
Status: Completed | Type: Observational
Sponsor: Comenius University (Other)
Collaborators: Pavol Jozef Safarik University (Other)
Responsible Party: Sponsor
Other Study IDs: EC UNM 115/2023
Record Dates: First submitted 2023-12-13; First posted 2024-01-25 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Stress Urinary Incontinence; Athletes
Keywords: Stress urinary incontinence; Athletes; Intravaginal pressure; Intra-abdominal pressure
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- sportwoman with high intensity of physical activity with stress urinary incontinence: High-intensity of regular physical activity at least three days per week, 90 minutes per day, for more than two years.
  Interventions: Diagnostic Test: intra-abdominal pressure with Femfit® device during (jumps on the ground, jumps on a trampoline, weightlifting, slow running, fast running
- sportwoman with high intensity of physical activity without stress urinary incontinence: High-intensity of regular physical activity at least three days per week, 90 minutes per day, for more than two years.
  Interventions: Diagnostic Test: intra-abdominal pressure with Femfit® device during (jumps on the ground, jumps on a trampoline, weightlifting, slow running, fast running

INTERVENTIONS:
Diagnostic Test: intra-abdominal pressure with Femfit® device during (jumps on the ground, jumps on a trampoline, weightlifting, slow running, fast running — Change in intravaginal and intra-abdominal pressure assessed by Femfit® , leakage of urine in grams assessed by inovative pad test during 5 sports activities.
  Other Names: intravaginal and intra-abdominal pressure with Femfit® device during (squeeeze, knack, rapid contractions, endurance contracions); inovative pad test during (jumps on the ground, jumps on a trampoline, weightlifting, slow running, fast running

SUMMARY:
To compare the impact of selected physical activities on pelvic floor and stress urinary incontinence in sportwoman.

DETAILED DESCRIPTION:
This is an observational comparative pilot study in which we will compare intravaginal and intra-abdominal pressure and an innovative pad test in 5 female athletes with stress urinary incontinence and 5 without incontinence.

ELIGIBILITY:
Inclusion criteria

* nulliparous women
* aged 18-35
* high-intensity physical activity
* performed sport at least three days per week, 90 minutes per day, for more than two years

Exclusion Criteria:

* handicapped sportswomen
* performance of various kinds of sport
* no regular sport activity
* performance of sports for less than two years
* after childbirth
* surgical treatment of gynaecological and urological illnesses
* urinary tract infection
* disease of respiratory tract
* not sufficiently completed questionnaires
* refusal to participate
* body mass index greater than 30 (BMI = m/h2, where m = body weight in kilograms and h = body height in metres)
* symptoms of overactive bladder

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: sportwoman with high intensity of physical activity with and without stress urinary incontinence
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
To measure intravaginal and intra-abdominal pressure with Femfit® device in sportwoman with and wihout Stress Urinary Incontinence. | During the performance of sporting activities up to 60 minutes.
  Intravaginal and intra-abdominal pressure will be measured in mmHg.

SECONDARY OUTCOMES:
To detect the amount of urine leakage by an innovative pad test in sportwoman. | During the performance of sporting activities up to 60 minutes.
  Leakage of urine will be measured by weight of pad in grams.
To detect the degree of urinary leakage by the International Consultation on Incontinence Questionnaire in sportwoman. | During the performance of sporting activities up to 60 minutes.
  Degree of leakage of urine will be measured by the International Consultation on Incontinence Questionnaire short form in score.

CONTACTS AND LOCATIONS:
Overall Officials: Magdaléna Hagovská, Dr., PhD, Study Director — Faculty of Medicine, PJ Safarik University, Kosice, Slovak Republic
Locations (1):
- Department of Urology, Jessenius Faculty of Medicine, Martin, Comenius University Bratislava, Slovak Republic, Martin, Slovakia, Slovakia

IPD SHARING:
Plan to Share IPD: No
On request

REFERENCES:
- [Background] Kruger JA, Dietz HP, Murphy BA. Pelvic floor function in elite nulliparous athletes. Ultrasound Obstet Gynecol. 2007 Jul;30(1):81-5. doi: 10.1002/uog.4027. PMID 17497753
- [Derived] Hagovska M, Bukova A, Svihra J. Measurement of the Vaginal Pressure Profile with the Femfit(R) and Leakage Events Using a Newly Developed Pad Test during Selected Sports Activities: A Pilot Study. Int Urogynecol J. 2025 Apr;36(4):789-797. doi: 10.1007/s00192-025-06051-y. Epub 2025 Jan 21. PMID 39836175